CLINICAL TRIAL: NCT00390169
Title: Randomized Controlled Trial Comparing Mindfulness-Based Stress Reduction (MBSR) to Supportive-Expressive Therapy (SET) on Psychological and Biological Outcomes in Breast Cancer Patients
Brief Title: Randomized Controlled Trial Comparing MBSR to SET in Breast Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Canadian Breast Cancer Research Alliance (Other)
Collaborators: British Columbia Cancer Agency (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 20444; CBCRA #017728
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-08

CONDITIONS: Breast Neoplasms
Keywords: breast neoplasms; stress; personality; psychology
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Behavioral: Mindfulness Meditation-Based Stress Reduction
Behavioral: Supportive-Expressive Group Therapy

SUMMARY:
This study will compare three standard treatment programs commonly offered to patients with breast cancer. The three programs being compared are 1) Mindfulness Meditation-Based Stress Reduction (MBSR), 2)Supportive- Expressive Group Therapy (SET), and 3) A one day stress-management seminar. The purpose of this study is to determine if these three treatments have different effects on psychological well-being, the immune system, and the amount of stress hormones in the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must be women diagnosed with Stage I, II, or III breast cancer within the previous 18 months, have completed all treatments with the exception of hormonal therapy at least three months previously, over the age of 18, and have a score of 13 or higher on the BSI-18. Previous meditation/yoga experience is allowed but will be recorded.

Exclusion Criteria:

* Participants must not have a concurrent DSM-IV diagnosis of psychosis, substance abuse, bipolar disorder, or active suicidality (as assessed by structured clinical interview), must not be currently using psychotropic medications (antipsychotics, antidepressants, anxiolytics), have a concurrent autoimmune disorder, or have participated previously in MBSR or SET group.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-10; Study Completion 2009-07

PRIMARY OUTCOMES:
Psychological:mood, stress, post-traumatic growth, social support, quality of life, spirituality
Physical:cortisol levels (stress hormone)

SECONDARY OUTCOMES:
emotional repression
personality
emotional suppression

CONTACTS AND LOCATIONS:
Overall Officials: Linda E Carlson, Ph.D, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

REFERENCES:
- [Background] Carlson LE, Garland SN. Impact of mindfulness-based stress reduction (MBSR) on sleep, mood, stress and fatigue symptoms in cancer outpatients. Int J Behav Med. 2005;12(4):278-85. doi: 10.1207/s15327558ijbm1204_9. PMID 16262547
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress and levels of cortisol, dehydroepiandrosterone sulfate (DHEAS) and melatonin in breast and prostate cancer outpatients. Psychoneuroendocrinology. 2004 May;29(4):448-74. doi: 10.1016/s0306-4530(03)00054-4. PMID 14749092
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress, and immune parameters in breast and prostate cancer outpatients. Psychosom Med. 2003 Jul-Aug;65(4):571-81. doi: 10.1097/01.psy.0000074003.35911.41. PMID 12883107
- [Derived] Carlson LE, Tamagawa R, Stephen J, Drysdale E, Zhong L, Speca M. Randomized-controlled trial of mindfulness-based cancer recovery versus supportive expressive group therapy among distressed breast cancer survivors (MINDSET): long-term follow-up results. Psychooncology. 2016 Jul;25(7):750-9. doi: 10.1002/pon.4150. Epub 2016 May 18. PMID 27193737
- [Derived] Carlson LE, Beattie TL, Giese-Davis J, Faris P, Tamagawa R, Fick LJ, Degelman ES, Speca M. Mindfulness-based cancer recovery and supportive-expressive therapy maintain telomere length relative to controls in distressed breast cancer survivors. Cancer. 2015 Feb 1;121(3):476-84. doi: 10.1002/cncr.29063. Epub 2014 Nov 3. PMID 25367403